CLINICAL TRIAL: NCT00707811
Title: Evaluation of ST2 and IL-33 for Risk Stratification and Diagnosis in Patients Presenting to the Emergency Department With Dyspnea
Brief Title: Evaluation of ST2 and IL-33 in Patients Presenting to the Emergency Department With Trouble Breathing
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Critical Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CCED08043
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Pulmonary Embolism; Pneumonia; Congestive Heart Failure
Keywords: Dyspnea; Shortness of Breath; Trouble Breathing; ST2; IL-33
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Pulmonary Embolism; Pneumonia; Heart Failure; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Trouble breathing (dyspnea) is a nonspecific symptom associated with many diseases such as chronic obstructive pulmonary disease (lung disorder in which the flow of air to the lungs is blocked), asthma, pneumonia, pulmonary hypertension (high blood pressure in the lungs), congestive heart failure (fluid build-up in the lungs because the heart is not pumping normally) and pulmonary embolism (blood clot in the lungs). The purpose of this study is to test two blood markers called ST2 and IL-33. Blood markers are proteins or other compounds in your blood that physicians use to diagnose different diseases and to determine what the course of an illness will be. In preliminary research studies, ST2 and IL-33 have been elevated in patients with a wide variety of diseases where the lungs are the primary organs involved. This research study will further investigate the ability of ST2 and IL-33 to predict the severity of disease and the possible use of ST2 and IL-33 in the diagnosis of various lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the Emergency Department with signs and symptoms of dyspnea (short of breath, tachypnea, hyperventilation, etc) within the last 24 hours
* Normal cardiac output as measured by noninvasive bioimpedance
* Greater than or equal to 18 years of age
* Patient or legal representative willing and able to provide informed consent and comply with study procedures

Exclusion Criteria:

* ECG changes diagnostic of acute myocardial ischemia/infarction
* Ischemic chest pain within the prior 24 hours by history
* Obvious chest trauma

Exclusion Criteria for Blood Draw:

* A history of congestive heart failure and a BNP > 500pg/mL (or NTproBNP > 900pg/mL) if obtained by the treating physician
* Treating physician suspects patient has new onset congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Cleveland Clinic Emergency Department with signs and/or symptoms of dyspnea (trouble breathing)
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Any cause of mortality | 180 days

SECONDARY OUTCOMES:
Rehospitalization of a pulmonary etiology and/or significant lung morbidity (transplant, intubation, ARDS, pneumonia, pulmonary hypertension, etc) | 180 days
Mortality with a pulmonary specific etiology | 180 days
Any cause morbidity | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Benoit, BS, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Lloyd CM, Hessel EM. Functions of T cells in asthma: more than just T(H)2 cells. Nat Rev Immunol. 2010 Dec;10(12):838-48. doi: 10.1038/nri2870. Epub 2010 Nov 9. PMID 21060320